CLINICAL TRIAL: NCT00354562
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of ABT-751 in Combination With Docetaxel Versus Docetaxel Alone in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Phase 2 Study Evaluating ABT-751 in Combination With Taxotere in Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Helen Eliopoulos, MD, Global Project Head, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M05-782; 2006-002838-38 (EudraCT Number)
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-09

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Lung Cancer; Non-Small Cell Lung Cancer; NSCLC; ABT-751; docetaxel; Taxotere
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — ABT751; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Docetaxel + ABT-751
  Interventions: Drug: ABT-751; Drug: Docetaxel
- B (Placebo Comparator): Docetaxel + placebo
  Interventions: Drug: Placebo; Drug: Docetaxel

INTERVENTIONS:
Drug: ABT-751 — 200mg ABT-751 daily for 14 days every 21 days
  Arms: A
Drug: Placebo — Placebo daily for 14 days every 21 days
  Arms: B
Drug: Docetaxel — Standard Docetaxel every 21 days
  Other Names: Taxotere

SUMMARY:
To determine the efficacy of ABT-751 when administered in combination with standard docetaxel in subjects with advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented NSCLC
* Locally advanced (Stage III) or metastatic (Stage IV) NSCLC
* Only one prior anti-tumor treatment regimen in the non-curative setting (i.e., 2nd-line therapy)
* Only one prior anti-tumor treatment regimen in the curative setting
* Progressive disease following the previous anti-tumor treatment regimen
* Measurable disease by RECIST criteria
* Brain metastasis must be stable and well-controlled

ECOG performance score 0-2All anti-tumor therapy discontinued at least 3 weeks prior to study entryAll adverse events from prior treatment are resolved or stableAdequate hematologic, renal, and hepatic functionFemales must not be pregnantWilling to take adequate measures to prevent pregnancyLife expectancy of at least 3 monthsAble to complete the Quality of Life questionnaireVoluntarily signed informed consent

* Only one prior anti-tumor treatment regimen in the curative setting
* Progressive disease following the previous anti-tumor treatment regimen
* Measurable disease by RECIST criteria
* Brain metastasis must be stable and well-controlled
* ECOG performance score 0-2
* All anti-tumor therapy discontinued at least 3 weeks prior to study entry
* All adverse events from prior treatment are resolved or stable
* Adequate hematologic, renal, and hepatic function
* Females must not be pregnant
* Willing to take adequate measures to prevent pregnancy
* Life expectancy of at least 3 months
* Able to complete the Quality of Life questionnaire
* Voluntarily signed informed consent

Exclusion Criteria:

* Greater that Grade 1 neurological findings
* Allergy to sulfa medications
* Previous treatment with ABT-751 or docetaxel
* Receipt of more than one investigational agent for NSCLC
* Significant weight loss (>10%) within 6 weeks of study entry
* Glucose-6-phosphate dehydrogenase deficiency or porphyria
* Significant systemic disease that would adversely affect participation
* Class 3-4 New York Heart Association classification status
* Other cancers except in situ carcinoma of the cervix, basal or squamous cell skin cancer, or any other cancer considered adequately treated and cured by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | Subjects may remain on study until disease progression

SECONDARY OUTCOMES:
Overall Survival | Subject may remain on study until disease progression
Response Rate | Subject may remain on study until disease progression
Time-to-Progression (TTP) | Subject may remain on study until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Helen Eliopoulos, MD, Study Director — Abbott
Locations (32):
- United States (13):
  - Site Ref # / Investigator 3572, Birmingham, Alabama
  - Site Ref # / Investigator 4771, Burbank, California
  - Site Ref # / Investigator 3574, Orange, California
  - Site Ref # / Investigator 3567, Rancho Mirage, California
  - Site Ref # / Investigator 3512, Gurnee, Illinois
  - Site Ref # / Investigator 3565, Hackensack, New Jersey
  - Site Ref # / Investigator 3569, Buffalo, New York
  - Site Ref # / Investigator 3511, Cleveland, Ohio
  - Site Ref # / Investigator 5237, Ravenna, Ohio
  - Site Ref # / Investigator 3551, Crossville, Tennessee
  - Site Ref # / Investigator 3549, Knoxville, Tennessee
  - Site Ref # / Investigator 3571, Nashville, Tennessee
  - Site Ref # / Investigator 3510, Weston, Wisconsin
- Canada (7):
  - Site Ref # / Investigator 3563, Sydney, Nova Scotia
  - Site Ref # / Investigator 3559, Barrie, Ontario
  - Site Ref # / Investigator 3561, Greater Sudbury, Ontario
  - Site Ref # / Investigator 3560, Greenfield Park, Quebec
  - Site Ref # / Investigator 3562, Montreal, Quebec
  - Site Ref # / Investigator 2222, Montreal, Quebec
  - Site Ref # / Investigator 3558, Regina, Saskatchewan
- Ireland (5):
  - Site Ref # / Investigator 5097, Cork
  - Site Ref # / Investigator 4971, Dublin
  - Site Ref # / Investigator 4986, Dublin
  - Site Ref # / Investigator 4999, Dublin
  - Site Ref # / Investigator 5158, Dublin
- United Kingdom (7):
  - Site Ref # / Investigator 5259, Belfast
  - Site Ref # / Investigator 5270, East Barming
  - Site Ref # / Investigator 5271, Edinburgh
  - Site Ref # / Investigator 5017, Glasgow
  - Site Ref # / Investigator 5274, Hull
  - Site Ref # / Investigator 5273, Surrey
  - Site Ref # / Investigator 5268, Surrey